CLINICAL TRIAL: NCT00556179
Title: Local, National (Brazil), Multicentric, Open, Non-Controlled, Phase IV, Study of Lactoserum (Dermacyd Femina®), in Women at Reproductive Age, to Prevent Recurrence of Bacterial Vaginosis, During Three Months, After Standard Treatment With Metronidazole.
Brief Title: Lactoserum (Dermacyd Femina®) and Prevention of Recurrence of Bacterial Vaginosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LACTO_L_02399
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — lactoserum

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lactoserum (Dermacyd Femina®)

INTERVENTIONS:
Drug: Lactoserum (Dermacyd Femina®) — Once a day during three months

SUMMARY:
The purpose of this study is to demonstrate if the use of Dermacyd can avoid the recurrence of bacterial vaginosis after three months of the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age
* Confirmed cure of bacterial vaginosis after treatment with oral metronidazole.
* Vaginal bacterioscopic examination negative for candida and trichomonas.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Allergy to dermacyd

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence of bacterial vaginosis after three months of treatment. | Three months

SECONDARY OUTCOMES:
Quality of life | Three months
Vaginal Candidiasis | Three months
AE, particularly genital irritation (tolerability use of dermacyd) | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis, São Paulo, São Paulo, Brazil